CLINICAL TRIAL: NCT03978416
Title: Development of Novel Behavioral Intervention for Sustainable Weight Loss in Hispanic Adults With Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to the SARS-CoV-2 pandemic. Aim 1 was completed.
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Maria Carlota Dao, Scientist, Tufts University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13352
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Hispanic / Latino; Older adults; Eating habits
MeSH Terms: conditions — Obesity; Weight Loss; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A prototype bilingual English-Spanish lifestyle intervention for weight reduction will be created. The prototype will then be iteratively refined during a series of short-term tests (two tests lasting 4 weeks, followed by a final test lasting 12 weeks) of intervention delivery. In these interventions, % weight loss, % drop-out, and safety benchmarks will be monitored. Participant-reported barriers to adherence identified during group meetings and exit interviews will be targets for improvement in successive iterations.
Masking Description: The purpose of this project is to develop a lifestyle intervention for weight loss by conducting three pilot studies where small groups of participants undergo progressively developed versions of the intervention. There will not be masking as both subjects and investigators will be aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focus groups (No Intervention): Information on practical and cultural barriers and promoters of successful weight management will be collected through focus groups. This will include include food access, dietary patterns, physical activity, time and financial constraints, and additional psychosocial and cultural factors.
  A total of 30 participants will be recruited for the focus groups.
- Pilot behavioral intervention (Experimental): A prototype bilingual English-Spanish lifestyle intervention for weight reduction will be created. The prototype will then be iteratively refined during a series of short-term tests with 5 participants per test (two tests lasting 4 weeks, followed by a final test lasting 12 weeks) of intervention delivery.
  Interventions: Behavioral: Healthy Weight for Living for Hispanics

INTERVENTIONS:
Behavioral: Healthy Weight for Living for Hispanics — The Healthy Weight for Living (HWL) intervention, previously developed at the Energy Metabolism Laboratory (HNRCA), is broadly informed by the same behavior change theories as other interventions. For example, it also recognizes individual and environmental factors as potential areas to support behavior change for weight regulation, and provides practical tools for facilitating new habits. However, the HWL places greater emphasis on the role of biology in influencing eating behavior, giving a central role to hunger and food cravings as modulators of eating behavior. Therefore, HWL does not emphasize self-monitoring food intake and does not require increasing physical activity for effectiveness. The new intervention also targets autonomous motivation and prioritizes ease of implementation.
  Information from focus groups and sequential pilots will be used to develop a culturally tailored prototype version of Healthy Weight for Living that is acceptable for Hispanic older adults.
  Arms: Pilot behavioral intervention

SUMMARY:
There are great disparities in the prevalence of obesity and chronic disease in different sociodemographic groups. US Hispanic adults, in particular, have a higher prevalence of obesity and chronic diseases than non-Hispanic whites. Population aging is also a major contributing factor to the high prevalence of chronic disease, and Hispanics already make up approximately 10% of the older population. Therefore, preventive measures are needed to reduce the burden of chronic disease risks for Hispanics. Current lifestyle interventions for weight management have been particularly ineffective in this population.

The purpose of this pilot project is to develop a novel tailored lifestyle intervention for use by Hispanic older adults with obesity. The Healthy Weight for Living intervention has been validated among adults with mixed racial/ethnic backgrounds and has achieved clinically impactful weight-loss. Its design features make it particularly suitable for use in populations with low adherence to traditional interventions, including no requirement for daily food logging and no increase in physical activity.

The final product of this project will be a culturally adapted prototype intervention in Hispanic older adults that accounts for cultural heterogeneity. This work has direct relevance to reducing health disparities and the burden of obesity-associated chronic disease in a particularly at-risk population.

DETAILED DESCRIPTION:
The scientific premise of this project is that appropriately tailored lifestyle interventions for weight loss can achieve clinically impactful weight loss in Hispanic adults with obesity. Older adults will be the focus, recognizing that requirements for tailoring may vary according to age group. Given that older adults have a higher risk of chronic diseases caused by obesity, there is a great need to focus on factors that disproportionately affect older Hispanic adults. The objective of this project is to tailor a validated lifestyle intervention developed and used by our team in ethnically mixed populations to older Hispanic adults with obesity. This novel intervention does not require food logging or a large increase in physical activity to achieve weight loss, making it more acceptable to population groups with low adherence to traditional interventions. The long-term goal of this work is to create an effective, culturally acceptable, sustainable, and scalable lifestyle weight management program for routine use in Hispanic adults with obesity. Findings from this work will be directly applicable to future community interventions and will be relevant for public health measures in this at-risk population.

The specific aims are:

Aim 1: To conduct focus groups in Hispanic older adults with obesity to identify factors that can be addressed in the tailored intervention. Information will be collected on practical and cultural barriers and promoters of successful weight management, including food access, dietary patterns, physical activity, time and financial constraints, and additional psychosocial and cultural factors.

Hypothesis 1: Malleable dietary and psychosocial targets for weight loss and weight loss maintenance can be identified, including factors such as food cravings, hunger and disinhibited eating that have been shown to be effective targets in other population groups.

Aim 2: To conduct a pilot behavioral intervention of an initially adapted program in Hispanic older adults with obesity. A prototype bilingual English-Spanish lifestyle intervention for weight reduction will be created. The prototype will then be iteratively refined during a series of short-term tests (two tests lasting 4 weeks, followed by a final test lasting 12 weeks) of intervention delivery. In these interventions, % weight loss, % drop-out, and safety benchmarks will be monitored. Participant-reported barriers to adherence identified during group meetings and exit interviews will be targets for improvement in successive iterations.

Hypothesis 2: Successive refinement of the program will result in progressive improvements in mean % weight loss and participant retention.

The final products of this project will be: a) a prototype adapted intervention in older US adults of Hispanic background, accounting for cultural heterogeneity in this population; and b) identification of additional barriers that can be addressed in subsequent iterations of the intervention.

ELIGIBILITY:
INCLUSION CRITERIA:

Focus groups and Intervention:

1. Adult men and women older than 50 years.
2. Self-identifying as having Hispanic ethnicity, originating from Spanish-speaking Latin-American country.
3. BMI ≥30.0 kg/m2.

   Intervention only:
4. Willing to give informed consent.
5. All individuals wishing to participate in the intervention part of this study will be required to agree to inform their physician prior to enrollment and to notify the Tufts team if their physician recommends against weight loss for any reason. A physician's clearance form will be provided by Tufts to all participants wishing to enroll in the intervention. Participants will be required to obtain their physicians' signature and their physician will send the completed form to us. We will enroll them only after we have obtained a signed physician clearance form.
6. Willing to participate in a behavioral intervention for weight loss.

EXCLUSION CRITERIA:

Intervention only:

1. Self-reported weight loss >5 kg within past 6 months.
2. Diagnosed gastrointestinal conditions, including celiac disease.
3. Communicable or chronic diseases or medication use that would preclude safe and active study participation.
4. Pregnancy or anticipated pregnancy within the study,
5. Lactation, or giving birth within 6 months prior to enrollment.
6. Participation in other clinical trials.
7. Illiteracy.
8. Use of anti-obesity medications within the past year.
9. Being on any special diets that would prevent following recommendations made through the program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Weight change | Pilot 1 and 2: 4 weeks. Pilot 3: 12 weeks
  Change in weight from baseline to the end of the intervention period
Attendance to weekly group meetings | Pilot 1 and 2: 4 weeks. Pilot 3: 12 weeks
  Adherence will be measured as meeting attendance

SECONDARY OUTCOMES:
Change in blood pressure (systolic and diastolic) | Depending on pilot phase the time frame will be 4 weeks or 12 weeks
  Change in systolic and diastolic blood pressure from baseline to the end of the intervention period
Change in waist circumference | Depending on pilot phase the time frame will be 4 weeks or 12 weeks
  Change in waist circumference from baseline to the end of the intervention period
Change in hip circumference | Depending on pilot phase the time frame will be 4 weeks or 12 weeks
  Change in hip circumference from baseline to the end of the intervention period
Themes generated from qualitative data | Baseline, 4 weeks for pilot cycles 1 and 2, and 12 weeks for pilot cycle 3
  For the first phase of the study, focus groups will be analyzed and themes on eating behavior and barriers to successful weight management will be identified.
  For the intervention phase of the study, exit interviews will be completed at the end of each pilot cycle.
Financial well-being | Baseline
  Financial well-being questionnaire (4 items). Financial satisfaction (1 item) Financial difficulty (1 item) Financial control (1 item) Scores are standardized and summed to capture financial well-being. Higher scores indicate more financial well-being.
Dietary intake | Baseline
  NHANES Dietary Screener Questionnaire (DSQ, 26 items). The DSQ scoring algorithms developed at the National Cancer Institute will be used to calculate estimated intakes of food groups and certain nutrients: fruits and vegetables (cup equivalents), dairy (cup equivalents), added sugars (teaspoon equivalents), whole grains (ounce equivalents), and fiber (g).
  Source: https://epi.grants.cancer.gov/nhanes/dietscreen/scoring/current/#scoring
Dietary behavior | Baseline
  Latino Dietary Behaviors Questionnaire (LDBQ, 13 items)
  Possible scores:
  Health dietary changes score range: 0 to 19 Artificial sweeteners in drinks score range: 0 to 13 Number of meals per day score range: 0 to 6 Fat consumption score range: 0 to 9 Total LDBQ score range (sum of all items): 0 to 47 Lower scores indicate poorer dietary behaviors.
Perceived stress | Baseline
  Perceived Stress Scale 4 (PSS-4, 4 items) Score range: 0 to 16. Higher scores are correlated to more stress.
Eating behavior (hunger, satiety, cognitive restraint) | Baseline
  Three factor eating questionnaire (TFEQ, 51 items) Cognitive restraint score range: 0 to 21 Disinhibition score range: 0 to 16 Hunger score range: 0 to 14 Higher scores indicate higher degrees of the particular eating behavior.
Acculturation | Baseline
  Short Acculturation Scale for Hispanics (SASH, 12 items) Each item response is based on a five-point bipolar scale. Scores are calculated by taking the average rating across all items. Higher scores indicate higher acculturation.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dao MC, Yu Z, Maafs-Rodriguez A, Moser B, Cuevas AG, Economos CD, Roberts SB. Perceived intrinsic, social, and environmental barriers for weight management in older Hispanic/Latino adults with obesity. Obes Sci Pract. 2022 Aug 31;9(2):145-157. doi: 10.1002/osp4.631. eCollection 2023 Apr. PMID 37034568